CLINICAL TRIAL: NCT02808858
Title: Rete Italiana Dei Registri Regionali Delle Sindromi Mielodisplastiche (MDS)
Brief Title: Italian Network MDS Registry
Acronym: FISM_registry
Status: Recruiting | Type: Observational
Sponsor: Fondazione Italiana Sindromi Mielodisplastiche-ETS (Other)
Responsible Party: Sponsor
Other Study IDs: Rete italiana registri MDS
Record Dates: First submitted 2016-05-18; First posted 2016-06-22 (Estimated); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Myelodysplastic-Myeloproliferative Diseases
Keywords: MDS; Myelodisplastic Syndrome
MeSH Terms: conditions — Myelodysplastic-Myeloproliferative Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Epidemiological data collection of adult patients affected by myelodysplastic syndrome (MDS) newly diagnosed.

DETAILED DESCRIPTION:
Development of an Italian regional registries MDS network using the same electronic case report form for data storage, with the following broad aims:

* Ability to aggregate and process anonymous epidemiological data collected by individual regional registers;
* Ability to aggregate the available data with those of other international registries existing.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of MDS

Exclusion Criteria:

* Patient who refuse the signature of informed consent

Ages: 18 Years to 106 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with new diagnosis of MDS
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-06 (Actual); Study Completion 2032-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of MDS diagnosis | 6 years
  Number of new cases every 100.000 person/year
Overall Response rate | 6 years
  Proportion of CR or PR after each line of treatment in term of erythroid, platelet and granulocyte response
Prevalence of MDS | 6 years
  Number of cases every 100.000 person
Overall survival | 6 years
  Time between MDS diagnosis and death due to any causes
Progression free survival | 6 years
  Time between MDS diagnosis and relapse/ progression or death due to any causes
Progression to AML | 6 years
  Time between MDS diagnosis and Progression to AML or death due to any causes

CONTACTS AND LOCATIONS:
Locations (20):
- Italy (20):
  - Ematologia, AO SS. Antonio e Biagio, Alessandria, AL
  - Clinica di Ematologia, AOU Ospedale di Torrette, Ancona, AN
  - U.O. Clinica Medicina Interna, IRCCS San Martino IST, Genova, GE
  - Struttura Cattedra di Ematologia e CTMO, AOU di Parma, Parma, PR
  - Ematologia e Centro Trapianti, Centro di Riferimento Oncologico della Basilicata, Rionero in Vulture, PZ
  - FPO - IRCCS di Candiolo, Candiolo, Torino
  - S.C.D.U. Ematologia e Terapie cellulari, Ospedale Mauriziano, Torino, TO
  - Ospedale Cardinal Massaia, Asti
  - Ematologia AOU Policlinico di Bari, Bari
  - Istituto di Ematologia e Oncologia Medica, Policlinico S.Orsola, Bologna
  - Ematologia- Ospedale Businco, Cagliari
  - Ospedale Maggiore, Chieri
  - Cattedra di Ematologia Policlino Careggi, Florence
  - Dipartimento Emato-Oncologia AOU San Martino Genova, Genova
  - Medicina interna II Divisione di Ematologia Ospedale S.Luigi Gonzaga, Orbassano
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliera Perugia, Perugia
  - AOU San Salvatore, Pesaro
  - Ospedale San Giovanbni Battista-Molinette, Torino
  - Divisione di Ematologia-Ospedale Cardinale Panico, Tricase

IPD SHARING:
Plan to Share IPD: No